CLINICAL TRIAL: NCT07110883
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Profiles, and Preliminary Efficacy of SYS6023 in Patients With Advanced Solid Tumors
Brief Title: A Clinical Study of SYS6023 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYS6023-001
Record Dates: First submitted 2025-07-14; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: All participants receive the same treatment, and there is no comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Dose-escalation group (Experimental): Patients with advanced solid tumors receiving SYS6023 treatment at doses ranging from 0.5 mg/kg to 6.5 mg/kg.
  Interventions: Drug: SYS6023
- Cohort-expansion A group (Experimental): Patients with Human Epidermal Growth Factor Receptor 3-positive(HER3+) / Hormone (estrogen and/or progesterone) receptor (HR)-positive (HR+)/ Human Epidermal Growth Factor Receptor 3-negative (HER2-) breast cancer receiving the recommended dose of SYS6023 treatment.
  Interventions: Drug: SYS6023
- Cohort-expansion B group (Experimental): Patients with EGFR-positive non-small cell lung cancer receiving the recommended dose of SYS6023 treatment.
  Interventions: Drug: SYS6023
- Cohort-expansion C group (Experimental): Patients with HER3+/HER2+ breast cancer receiving the recommended dose of SYS6023 treatment.
  Interventions: Drug: SYS6023
- Cohort-expansion D group (Experimental): Patients with HER3+ platinum-resistant and recurrent ovarian cancer receiving the recommended dose of SYS6023 treatment.
  Interventions: Drug: SYS6023
- Cohort-expansion E group (Experimental): Patients with locally advanced or metastatic non-small cell lung cancer positive for driver genes other than EGFR receiving the recommended dose of SYS6023 treatment.
  Interventions: Drug: SYS6023
- Cohort-expansion F group (Experimental): Patients with other types of HER3+ advanced solid tumors receiving the recommended dose of SYS6023 treatment.
  Interventions: Drug: SYS6023

INTERVENTIONS:
Drug: SYS6023 — SYS6023 is a novel antibody-drug conjugate (ADC) targeting HER3, administered via intravenous infusion.

SUMMARY:
This is an open-label, dose-escalation and cohort-expansion, multicenter Phase I study involving participants with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, dose-escalation and cohort-expansion, multicenter Phase I study involving participants with advanced solid tumors.

The study aims to evaluate the safety/tolerability, pharmacokinetics, and preliminary efficacy of SYS6023 in participants with advanced solid tumors.

The eligible subjects will receive intravenous infusion of SYS6023 on the first day of each cycle, with each treatment cycle lasting 3 weeks, until disease progression, intolerable toxicity, initiation of a new anti-tumor treatment, withdrawal of informed consent, loss to follow-up, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Histologically and/or cytologically confirmed locally advanced unresectable or metastatic malignant solid tumor;
3. Sufficient archived or fresh tumor tissue samples must be provided for HER3 testing, among others;
4. Medical documentation must be provided before the first dose to clarify the following molecular typing information: HER2, HR receptor (including estrogen receptor (ER) and progesterone receptor (PR) ) expression for breast cancer participants, and Epidermal Growth Factor Receptor (EGFR) mutation, Anaplastic Lymphoma Kinase (ALK) fusion, ROS Proto-Oncogene 1, receptor tyrosine kinase (ROS1) fusion, B-Raf Proto-Oncogene, serine/threonine kinase (BRAF) V600 mutation, Neurotrophic Tyrosine Receptor Kinase (NTRK) fusion, Neurotrophic Tyrosine Receptor Kinase (RET) rearrangement, HER2 mutation, MET Proto-Oncogene（Met）exon14 skipping mutation, Met amplification, KRAS Proto-Oncogene, GTPase G12C（KRAS G12c） mutation status for non-small cell lung cancer (NSCLC) participants;
5. Depending on the trial phase, the following requirements must be met:

   * **Cohort Expansion Phase:**
   * **Cohort A:** HER3+ (by central lab), HR+/HER2- (HR+ defined as expressing estrogen receptor (ER), with or without progesterone receptor (PR) co-expression), locally advanced or metastatic breast cancer, previously treated with at least one line of systemic therapy including endocrine and CDK4/6 inhibitor treatment.
   * **Cohort B:** EGFR mutation-positive locally advanced or metastatic non-small cell lung cancer, previously treated with at least one line of systemic therapy, including EGFR Tyrosine Kinase Inhibitor (TKI) and platinum-based chemotherapy.
   * **Cohort C:** HER3+ (by central lab), HER2+, locally advanced or metastatic breast cancer, previously treated with at least two lines of anti-HER2 systemic therapy including trastuzumab, taxane, and T-DM1 or TKI.
   * **Cohort D:** HER3+ (by central lab), platinum-resistant recurrent ovarian cancer (defined as disease progression within >3 months and ≤6 months after last platinum-based chemotherapy for first-line, or within 6 months for second-line or higher lines of platinum-based chemotherapy), and non-platinum refractory (defined as disease progression within 4 weeks after last platinum-based chemotherapy).
   * **Cohort E:** Other driver gene-positive (e.g., ALK fusion, ROS1 fusion, BRAF V600 mutation, NTRK fusion, RET rearrangement, HER2 mutation, Met exon 14 skipping mutation, Met amplification, KRAS G12c mutation, etc.), locally advanced or metastatic non-small cell lung cancer, previously treated with corresponding targeted TKI therapy.
   * **Cohort F:** other HER3+ (by central lab) tumor types (including but not limited to triple negative breast cancer (TNBC), driver gene mutation-negative NSCLC, prostate cancer, etc.) which may potentially benefit from this treatment, or known NRG1 fusion tumors, both of which have previously treated with at least one line of systemic therapy.
6. At least one measurable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST)1.1 criteria;
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1;
8. Expected survival of at least 3 months;
9. Adequate organ function, with laboratory test results meeting the following criteria (no blood transfusions, Erythropoietin, Erythropoietin, or other medical support treatments within 14 days before testing):

   * Absolute Neutrophil Count (ANC) ≥ 1.5 × 10^9/L
   * Platelet ≥ 100 × 10^9/L
   * Hemoglobin (Hb) ≥ 90 g/L
   * Total Bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), or TBIL ≤ 3 × ULN for participants with liver metastasis, liver cancer, or Gilbert's syndrome
   * Aspartate Aminotransferase (ALT) and Alanine Aminotransferase (AST) ≤ 2.5 × ULN, or ALT and AST ≤ 5 × ULN for participants with liver metastasis or liver cancer
   * Creatinine clearance (Ccr) > 50 mL/min (calculated using Cockcroft-Gault formula)
   * Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; International Normalized Ratio (INR) ≤ 1.5 × ULN
   * Left ventricular ejection fraction (LVEF) ≥ 50%
10. Fertile participants (both male and female) must agree to use reliable contraceptive methods (hormonal contraception, barrier methods, or abstinence) during the trial and for at least 6 months after the last dose; female participants of childbearing potential must have a negative blood pregnancy test within 7 days before enrollment;
11. Fully understand the clinical trial and voluntarily sign a written informed consent.

Exclusion Criteria:

* 1. Known symptomatic central nervous system or meningeal metastases, or other evidence of uncontrolled central nervous system or meningeal metastases as judged by the investigator; stable central nervous system or meningeal metastases are allowed; 2. Previous treatment with HER3-targeting ADC; 3. Adverse reactions from previous anti-tumor treatments that have not recovered to ≤ Grade 1 according to CTCAE 5.0 (excluding toxicities deemed not a safety risk by the investigator, such as alopecia); 4. Receipt of antibody-based macromolecule therapy, definitive radiotherapy, immunotherapy within 28 days before the first dose, or chemotherapy, small molecule targeted therapy, palliative radiotherapy, hormone therapy, or traditional Chinese medicine with anti-tumor indication effects within 14 days or 5 half-lives (whichever is longer) before the first dose; 5. Concurrent participation in another clinical trial, unless it is an observational (non-interventional) clinical trial or in the follow-up period of an interventional trial; 6. Receipt of major surgery or invasive intervention within 28 days before the first dose; 7. Known severe allergic reactions to the investigational intervention or any of its components or excipients; 8. Active bacterial, fungal, or viral infection requiring intravenous antibacterial, antifungal, or antiviral treatment before the first dose. Participants receiving prophylactic infection treatment without active infection symptoms may be considered for inclusion; 9. Uncontrolled serous cavity effusion (e.g., pleural effusion, ascites, pericardial effusion, etc.) requiring frequent drainage or medical intervention within 7 days before the first dose, excluding exfoliation cytology of exudate; 10. History of immunodeficiency, including Human immunodeficiency virus (HIV) antibody positivity; 11. Hepatitis B Surface Antigen (HBsAg) positive with Hepatitis B Virus (HBV)-DNA higher than the lower limit of detection or 1000 copies/mL (500 IU/mL) (whichever is lower), Hepatitis C virus (HCV) antibody positive with HCV-RNA higher than the lower limit of detection or 1000 copies/mL (whichever is lower); 12. Severe cardiovascular disease history, including but not limited to:
* Severe cardiac arrhythmia or conduction abnormality requiring clinical intervention, such as ventricular arrhythmia, grade II-III atrioventricular block, etc.;
* Average QT interval corrected by Fridericia's formula (QTcF) > 450 ms on three resting 12-lead Electrocardiogram;
* Acute coronary syndrome, congestive heart failure, stroke, or other grade 3 or higher cardiovascular events within 6 months before the first dose;
* New York Heart Association (NYHA) classification ≥ Class II;
* Any factors increasing the risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death in a first-degree relatives under 40 years old, concomitant use of drugs known to prolong QT interval;
* Uncontrolled hypertension (screening systolic BP ≥ 160 mmHg and/or diastolic Blood Pressure (BP) ≥ 100 mmHg); 13. Drug-induced colitis, or history of hormone-requiring interstitial lung disease/pneumonitis or current suspicion of interstitial lung disease/pneumonitis on screening imaging; 14. Evidence of gastrointestinal bleeding or perforation risk, or pyloric obstruction, persistent recurrent vomiting (defined as vomiting ≥ 3 times within 24 hours), deemed unsuitable for inclusion by the investigator; 15. Use of or need for strong Recombinant Human CYP3A4 Enzyme (CYP3A4) inducers or inhibitors, Organic Anion Transporting Polypeptides 1B1 (OATP1B1) or Organic Anion Transporting Polypeptides 1B3 (OATP1B3) inhibitors within 5 half-lives before the first dose or during the study; 16. Current psychiatric disorder affecting compliance; 17. Exclusion of those on long-term immunosuppressive therapy or requiring daily systemic steroid treatment, except for topical glucocorticoid treatment via nasal, inhalation, or other routes; 18. Pregnant or breastfeeding women; 19. Other reasons deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose-limiting toxicity (DLT) | At the end of Cyecle 1 (each cycle is 21 days).
  DLTs are quantified using Common Terminology Criteria for Adverse Events（CTCAE）5.0
Number of Participants Reporting Adverse Events (AEs) and Serious Adverse Events (SAEs) (according to NCI-CTCAE 5.0) | Baseline up to 28 days post last dose,. Up to approximately 2 years.
  AEs and SAEs are quantified using Common Terminology Criteria for Adverse Events（CTCAE） 5.0
Recommended Phase 2 Dose（RP2D） | Up to approximately 2 years
  The "Recommended Phase 2 Dose" (RP2D) refers to the optimal dosage of the drug identified during Phase 1 clinical trials, which is then suggested for use in Phase 2 trials. This dosage is chosen based on a balance of factors including safety, tolerability, pharmacokinetics (how the drug is absorbed, distributed, metabolized, and excreted in the body), and preliminary efficacy data.

SECONDARY OUTCOMES:
Area Under the Serum Concentration Time Curve ( AUC) | Up to approximately 4 years
  The serum concentrations were quantified using the IC-LC/MS assay.
Maximum Plasma Concentration( Cmax) | The serum concentrations were quantified using the IC-LC/MS assay.
  The serum concentrations were quantified using the IC-LC/MS assay.
Minimum Plasma Concentration ( Cmin) | Up to approximately 4 years
  The serum concentrations were quantified using the IC-LC/MS assay.
Time to Maximum Plasma Concentration (Tmax) | Up to approximately 4 years
  The serum concentrations were quantified using the IC-LC/MS assay.
Anti-Drug Antibody（ADA） | Up to approximately 4 years.
  The serum concentrations were quantified using the ELISA assay.
Overall response rate (ORR) | Up to approximately 4 years.
  ORR will be evaluated using RECIST v1.1.
Disease control rate (DCR) | Up to approximately 4 years.
  DCR will be evaluated using RECIST v1.1.
Duration of Response (DoR) | Up to approximately 4 years.
  DoR will be evaluated using RECIST v1.1.
Progression-Free-Survival (PFS) | Up to approximately 4 years.
  PFS will be evaluated using RECIST v1.1.
Overall survival (OS) | Up to approximately 4 years
  OS will be evaluated using RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, M.D., Study Chair — Shanghai Chest Hospital; Qingyuan Zhang, M.D., Study Chair — Affiliated Tumor Hospital of Harbin
Locations (2):
- China (2):
  - Affiliated Tumor Hospital of Harbin, Harbin, Heilongjiang
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality